CLINICAL TRIAL: NCT00602927
Title: Neural Substrates of Varenicline's (Chantix®) Efficacy for Smoking Cessation
Brief Title: Effects of Varenicline on Brain Activity During Nicotine Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Dr. Caryn Lerman, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 806623; GA30517A (Other: Pfizer); P50CA084718 (NIH)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Nicotine Dependence
Keywords: Varenicline, Imaging, fMRI
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Varenicline (Active Comparator)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Day 1 - Day 3 0.5mg once daily Day 4 - Day 7 0.5mg twice daily Day 8 - Day 13 1.0mg twice daily
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Participants will take placebo pills for 13 days using the same regimen as the varenicline study period.
  Arms: Placebo

SUMMARY:
This project aims to define mechanisms through which varenicline might be an effective smoking cessation medication.

DETAILED DESCRIPTION:
Thirty treatment seeking smokers will be recruited to complete a 40-day within-subject (cross-over), double-blind study that will assess effects of varenicline on brain activation while performing certain tasks. Prior to beginning the study, participants will complete an health and physical screening to determine final eligibility. Following a medication run-up and a 3.5 day abstinence period, participants will complete study period 1 (an fMRI scan while performing attention, working memory and emotion tasks). After a 14 to 21-day washout period the study procedures will be repeated with placebo (order of study medication counterbalanced). After completion of both study periods, all participants will be offered a 13-week quit smoking program with varenicline.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-seeking smokers between the ages of 18 and 65, that smoke at least 10 cigarettes/day for at least the past 6 months
2. Provide a baseline CO (carbon monoxide) reading of >10ppm
3. Provide written informed consent and are fluent, English-speaking
4. Weight of equal to or less than 300 lbs

Exclusion Criteria:

Smoking Behavior

1. Use of chewing tobacco, snuff or cigars
2. Current enrollment or plans to enroll in another smoking cessation program in the next 5 months
3. Plan to use other nicotine substitutes or smoking cessation treatments in the next 5 months
4. Provide a baseline CO (carbon monoxide) reading ≤10 ppm

Alcohol/Drug Exclusion Criteria

1. History of substance abuse and/or currently receiving treatment for substance abuse
2. Current alcohol consumption that exceeds 25 standard drinks/week
3. A breath alcohol concentration reading ≥ 0.01 at the H&P (health & physical) screening or either of the lab sessions

Medication Exclusion Criteria

1. Prior use of Chantix
2. Current use or recent discontinuation (within last 14-days) of the following medications:

   1. Any form of smoking cessation medication
   2. Any form of anti-psychotic medications that includes:

      * antipsychotics,
      * atypical antipsychotics,
      * mood-stabilizers,
      * anti-depressants (tricyclic, SSRI, MAOI),
      * anti-panic agents,
      * anti-obsessive agents,
      * anti-anxiety agents, and
      * stimulants (e.g., Provigil, Ritalin)
      * herbal medications (St. John's Wort)
   3. Opioid medication for chronic pain
   4. Anti-coagulants
   5. Any heart medications
   6. Daily medication for asthma

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy, or lactating;
2. History or current diagnosis of psychosis, current major depression, bipolar disorder, ADHD, schizophrenia, or any Axis 1 disorder as identified by the MINI
3. Serious or unstable disease within the past 6 months (heart disease, HIV)
4. Diagnosis of cancer in the past 6 months or if successful treatment for cancer has not ended within the past 6 months
5. History of epilepsy or a seizure disorder
6. History or current diagnosis (last 6-months) of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of COPD (chronic obstructive pulmonary disease), cardiovascular disease (stroke, angina, coronary heart disease), heart attack in the last 6 months, uncontrolled hypertension (SBP>150 or DBP>90)
7. History of kidney and/or liver failure (including transplant)
8. History of head trauma or prior seizure; family history of a seizure disorder, brain (or central nervous system) tumor
9. Use of pacemakers, certain metallic implants, or presence of metal in the eye as contraindicated for MRI (magnetic resonance imaging);
10. Low or borderline intellectual functioning - determined by receiving a score <80 on the Shipley verbal IQ Test
11. Non-English speaking; determined at phone screen
12. History of claustrophobia (contraindicated for MRI) or color blindness (task requires color recognition); self-report at telephone screen
13. Being left-handed
14. Any fore-limb deformity
15. Wearing cochlear implant or bi-lateral hearing aids

General Exclusion

1. Any medical condition or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.
3. Any physical or visual impairment that may prevent the individual from using a computer keyboard or completing any study tasks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Tobacco Use Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Loughead J, Ray R, Wileyto EP, Ruparel K, Sanborn P, Siegel S, Gur RC, Lerman C. Effects of the alpha4beta2 partial agonist varenicline on brain activity and working memory in abstinent smokers. Biol Psychiatry. 2010 Apr 15;67(8):715-21. doi: 10.1016/j.biopsych.2010.01.016. Epub 2010 Mar 6. PMID 20207347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from mass media advertising in the greater Philadelphia area from November 2007 - June 2008.
Pre-assignment Details: All participants completed a 14 day wash-out period between the two study phases. They were instructed to resume their usual smoking behavior in this wash-out phase.
Groups:
- Placebo First, Then Varenicline; Varenicline First, Then Placebo: Days 1 - 3: 0.5 mg once a day orally Days 4 - 7: 0.5 mg twice a day orally Days 8 - 13: 1 mg twice a day orally
Period: Period 1: 13 Days
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 19 | 19
Completed | 15 | 14
Not Completed | 4 | 5
Not completed — Protocol Violation | 2 | 4
Not completed — MRI scanner technical issue | 1 | 0
Not completed — Time | 1 | 0
Not completed — Claustrophobia | 0 | 1
Period: Period 2: 14 Days
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 15 | 14
Completed | 15 | 12
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2
Period: Period 3: 13 Days
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 15 | 12
Completed | 13 | 9
Not Completed | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — MRI data quality | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.05 (13.32) | 39.79 (12.68) | 40.42 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percent Change BOLD Signal
Description: We calculated the percent BOLD signal change while performing the N-back task between the varenicline vs. placebo session. We subtracted BOLD signal observed during the 0-back condition from the BOLD signal observed during the 3-back condition (3back minus 0-back)We controlled for relevant co-variates such as sex, nicotine dependence level and education.
Time Frame: Day 13
Population: Participants who completed both study phases were included in the analyses (n=25). Additional participants (n=3) were excluded due to measurement artifact.
Measure: Mean (Standard Error); unit: BOLD Signal Change (3-back minus 0-back)
Groups:
- Placebo; Varenicline: Days 1 - 3: 0.5 mg once a day orally Days 4 - 7: 0.5 mg twice a day orally Days 8 - 13: 1 mg twice a day orally
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 22 | 22
BOLD Signal Change (3-back minus 0-back) | 0.48 (0.05) | 0.61 (0.03)

2. Secondary Outcome: Effect of Varenicline Treatment on Task Performance (N-back Correct Response Time)
Description: We examined the difference in correct reaction time on the N-back task between varenicline and placebo treatment. Models included terms for the main effect of treatment period (varenicline vs. placebo), memory load (0-back, 1-back, 2-back, 3-back) and covariates. We tested for interactions between nicotine dependence severity and treatment.
Time Frame: Day 13
Population: Participants who completed both study phases were included in the analysis. Other participants (n=3) were excluded due to measurement artifact.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 22 | 22
Milliseconds | 692.14 (128.57) | 637.99 (164.30)

ADVERSE EVENTS:
Time Frame: Day 13
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo First, Then Varenicline (N=19) | Varenicline First, Then Placebo (N=19)
Severe Lethargy (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No